CLINICAL TRIAL: NCT02176265
Title: Qvanteq Bioactive Coronary Stent System First in Man (FIM) Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qvanteq AG (Industry)
Collaborators: Cardialysis BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUEST I
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
Keywords: CAD; PCI; bioactive coronary stent; OCT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Qvanteq bioactive coronary stent system (Experimental): Open-label, single arm, non-randomized study
  Interventions: Device: Qvanteq bioactive coronary stent

INTERVENTIONS:
Device: Qvanteq bioactive coronary stent — PCI

SUMMARY:
Objective of this First in Man study is to assess feasibility and safety of Qvanteq's bioactive coronary stent for treatment of stable coronary artery disease patients with de novo coronary artery stenosis in native vessels.

The proprietary surface of Qvanteq's bioactive coronary stent improves the in-growth behavior of the stent in the treated vessel. In-vivo animal studies revealed fast in-growth (similar to BMS), which however is not resulting in excessive tissue overgrowth as observed in BMS but rather has an efficacy profile similar to drug-eluting stent (DES), meaning suppression of tissue overgrowth. This should reduce the risk of restenosis and thrombus formation despite the presence of a short term dual anti platelet therapy (DAPT). Furthermore, prolonged DAPT time as applied with current DES increases the bleeding risk of patients.

The study is a prospective, multicenter, open-label, single arm study; conducted in up to 6 cardiology centers in CH and NL. In total, approx. 35 patients will be enrolled. All patients will be treated with the Qvanteq's bioactive coronary stent. Clinical follow-up will occur at 1, 6 & 12 months post-stent implantation. All patients will undergo angiography assessment (QCA) and Optical Coherence Tomography investigation (OCT) at baseline and at 6 months follow-up. Baseline OCT should be performed after the successfully completed angiographic procedure (documentary OCT). 1 and 12 months clinical follow-ups are conducted via telephone.

Primary Angiographic endpoint is in-stent Late Lumen Loss at 6 months; assessed by off-line QCA. Primary OCT endpoint is mean neointimal thickness at 6 months; assessed by off-line OCT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Evidence of myocardial ischemia without elevated cardiac biomarkers (e.g. stable or unstable angina with stable haemodynamic condition, silent ischemia demonstrated by positive territorial functional study)
* The patient has a planned intervention of one single de novo lesion in one or two separate major epicardial territories (LAD, LCX, or RCA).
* The lesion must have a visually estimated diameter stenosis of ≥ 50% and < 100%
* Lesion length must be ≤16 mm
* The vessel size must be between 2.5 and 3.5 mm
* Written informed consent
* The patient agrees to the follow-up visits including angiographic follow-up and OCT control at 6 months

Key Exclusion Criteria:

* Evidence of ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of procedure.
* Patient suffered from stroke/TIA or myocardial infarction during the last 6 months
* LVEF <30%
* Platelet count <100,000 cells/mm3 or >400,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Known renal insufficiency (Creatinine clearance less than 30 mL/Min), or subject on dialysis, or acute kidney failure
* Patient undergoing planned surgery within 6 months with the necessity to stop ASA
* Patient requiring prolonged DAPT for other diagnoses (>1 month)
* History of bleeding diathesis or coagulopathy
* Patient requiring oral anticoagulation (Coumadin, NOAC)
* The patient is a recipient of a heart transplant
* Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel or cobalt-chromium
* Other medical illness (e.g. cancer, stroke with neurological deficiency) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy
* Female of child bearing potential (age <50 years and last menstruation within the last 12 months), who did not underwent tubal ligation, ovariectomy or hysterectomy.
* Previous CABG

Angiographic Exclusion Criteria:

* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
* Target lesion in left main stem.
* Target lesion involves a side branch > 2.0mm in diameter
* Aorto-ostial target lesion (within 3 mm of the aorta junction).
* Total occlusion or TIMI flow <3, prior to wire crossing
* The target vessel contains visible thrombus
* Restenotic lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
In-stent Late Lumen Loss (LLL) assessed by off-line QCA | At 6 months after stent implantation
Mean neointimal thickness assessed by off-line OCT analysis | At 6 months after stent implantation

SECONDARY OUTCOMES:
Acute lumen gain assessed by off-line QCA | At 6 months after stent implantation
In-segment Late Lumen Loss assessed by off-line QCA | At 6 months after stent implantation
Mean Lumen Diameter (MLD) assessed by off-line QCA | At 6 months after stent implantation
Diameter stenosis assessed by off-line QCA | At 6 months after stent implantation
Binary restenosis (diameter stenosis > = 50%) assessed by off-line QCA | At 6 months after stent implantation
Prolapse area/volume assessed by off-line OCT analysis | At baseline
Mean/minimal lumen diameter/area/volume assessed by off-line OCT analysis | At baseline and at 6 months after stent implantation
Mean/minimal stent diameter/area/volume assessed by off-line OCT analysis | At baseline and at 6 months after stent implantation
Stent symmetry assessed by off-line OCT analysis | At baseline and at 6 months after stent implantation
Stent expansion assessed by off-line OCT analysis | At baseline and at 6 months after stent implantation
Incomplete strut apposition assessed by off-line OCT analysis | At baseline and at 6 months after stent implantation
In-stent neointimal hyperplasia volume obstruction (%) assessed by off-line OCT analysis | At 6 months after stent implantation
Neointimal hyperplasia area/volume assessed by off-line OCT analysis | At 6 months after stent implantation
Mean/maximal thickness of the struts coverage assessed by off-line OCT analysis | At 6 months after stent implantation
Percentage number of covered struts assessed by off-line OCT analysis | At 6 months after stent implantation
Percentage of incomplete apposed struts assessed by off-line OCT analysis | At 6 months after stent implantation
Healing score assessed by off-line OCT analysis | At 6 months after stent implantation
Acute success (device and procedural) | At baseline
Device-oriented composite endpoints (cardiac death, MI not clearly attributable to a non-intervention vessel, clinically indicated target lesion revascularization) | At 1, 6 and 12 months after stent implantation
Myocardial infarction (Q-wave, Non q-wave) | At 1, 6 and 12 months after stent implantation
Clinically indicated revascularization of the target vessel | At 1, 6 and 12 months after stent implantation
Any revascularization | At 1, 6 and 12 months after stent implantation
Stent thrombosis according to ARC definitions | Up to 12 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD, Principal Investigator — Dep. of Cardiology, University Hospital Bern, Switzerland; Patrick W Serruys, Prof, Study Chair — Erasmus Medical Center, Thoraxcenter, Rotterdam, the Netherlands
Locations (6):
- Netherlands (2):
  - Thoraxcentrum Twente, Medisch Spectrum Twente, Enschede
  - Thoraxcenter Erasmus MC Universitair Medisch Centrum Rotterdam, Rotterdam
- Switzerland (4):
  - Universitätsklinik für Kardiologie Schweizer Herz- und Gefässzentrum Bern, Bern
  - Cardiologie interventionnelle HUG - Hôpitaux Universitaires de Genève, Geneva
  - HerzKlinik Hirslanden, Zurich
  - Stadtspital Triemli Zürich Klinik für Kardiologie, Zurich

REFERENCES:
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Raber L, Magro M, Stefanini GG, Kalesan B, van Domburg RT, Onuma Y, Wenaweser P, Daemen J, Meier B, Juni P, Serruys PW, Windecker S. Very late coronary stent thrombosis of a newer-generation everolimus-eluting stent compared with early-generation drug-eluting stents: a prospective cohort study. Circulation. 2012 Mar 6;125(9):1110-21. doi: 10.1161/CIRCULATIONAHA.111.058560. Epub 2012 Feb 1. PMID 22302840
- [Background] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578
- [Background] Ndrepepa G, Schuster T, Hadamitzky M, Byrne RA, Mehilli J, Neumann FJ, Richardt G, Schulz S, Laugwitz KL, Massberg S, Schomig A, Kastrati A. Validation of the Bleeding Academic Research Consortium definition of bleeding in patients with coronary artery disease undergoing percutaneous coronary intervention. Circulation. 2012 Mar 20;125(11):1424-31. doi: 10.1161/CIRCULATIONAHA.111.060871. Epub 2012 Feb 17. PMID 22344040
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Guagliumi G, Sirbu V, Musumeci G, Gerber R, Biondi-Zoccai G, Ikejima H, Ladich E, Lortkipanidze N, Matiashvili A, Valsecchi O, Virmani R, Stone GW. Examination of the in vivo mechanisms of late drug-eluting stent thrombosis: findings from optical coherence tomography and intravascular ultrasound imaging. JACC Cardiovasc Interv. 2012 Jan;5(1):12-20. doi: 10.1016/j.jcin.2011.09.018. PMID 22230145
- [Background] Pfisterer M, Brunner-La Rocca HP, Buser PT, Rickenbacher P, Hunziker P, Mueller C, Jeger R, Bader F, Osswald S, Kaiser C; BASKET-LATE Investigators. Late clinical events after clopidogrel discontinuation may limit the benefit of drug-eluting stents: an observational study of drug-eluting versus bare-metal stents. J Am Coll Cardiol. 2006 Dec 19;48(12):2584-91. doi: 10.1016/j.jacc.2006.10.026. Epub 2006 Nov 2. PMID 17174201
- [Background] Eisenstein EL, Anstrom KJ, Kong DF, Shaw LK, Tuttle RH, Mark DB, Kramer JM, Harrington RA, Matchar DB, Kandzari DE, Peterson ED, Schulman KA, Califf RM. Clopidogrel use and long-term clinical outcomes after drug-eluting stent implantation. JAMA. 2007 Jan 10;297(2):159-68. doi: 10.1001/jama.297.2.joc60179. Epub 2006 Dec 5. PMID 17148711
- [Background] Park SJ, Park DW, Kim YH, Kang SJ, Lee SW, Lee CW, Han KH, Park SW, Yun SC, Lee SG, Rha SW, Seong IW, Jeong MH, Hur SH, Lee NH, Yoon J, Yang JY, Lee BK, Choi YJ, Chung WS, Lim DS, Cheong SS, Kim KS, Chae JK, Nah DY, Jeon DS, Seung KB, Jang JS, Park HS, Lee K. Duration of dual antiplatelet therapy after implantation of drug-eluting stents. N Engl J Med. 2010 Apr 15;362(15):1374-82. doi: 10.1056/NEJMoa1001266. Epub 2010 Mar 15. PMID 20231231
- [Background] Gwon HC, Hahn JY, Park KW, Song YB, Chae IH, Lim DS, Han KR, Choi JH, Choi SH, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Jang Y, Kim HS. Six-month versus 12-month dual antiplatelet therapy after implantation of drug-eluting stents: the Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting (EXCELLENT) randomized, multicenter study. Circulation. 2012 Jan 24;125(3):505-13. doi: 10.1161/CIRCULATIONAHA.111.059022. Epub 2011 Dec 16. PMID 22179532
- [Background] Valgimigli M, Campo G, Monti M, Vranckx P, Percoco G, Tumscitz C, Castriota F, Colombo F, Tebaldi M, Fuca G, Kubbajeh M, Cangiano E, Minarelli M, Scalone A, Cavazza C, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R; Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia Study (PRODIGY) Investigators. Short- versus long-term duration of dual-antiplatelet therapy after coronary stenting: a randomized multicenter trial. Circulation. 2012 Apr 24;125(16):2015-26. doi: 10.1161/CIRCULATIONAHA.111.071589. Epub 2012 Mar 21. PMID 22438530
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Soehnlein O, Wantha S, Simsekyilmaz S, Doring Y, Megens RT, Mause SF, Drechsler M, Smeets R, Weinandy S, Schreiber F, Gries T, Jockenhoevel S, Moller M, Vijayan S, van Zandvoort MA, Agerberth B, Pham CT, Gallo RL, Hackeng TM, Liehn EA, Zernecke A, Klee D, Weber C. Neutrophil-derived cathelicidin protects from neointimal hyperplasia. Sci Transl Med. 2011 Oct 5;3(103):103ra98. doi: 10.1126/scitranslmed.3002531. PMID 21974936